CLINICAL TRIAL: NCT02105246
Title: Improving Delivery of Patient-Centered Cardiac Rehabilitation
Brief Title: The Healthy Heart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHR13-10887
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Cardiac Rehabilitation
Keywords: cardiovascular disease; cardiac rehabilitation; secondary prevention; comparative effectiveness; 6 minute walk test
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based (Experimental): Referral to a home-based cardiac rehabilitation program (intervention).
  Interventions: Behavioral: Referral to center-based cardiac rehab
- Center-based (Active Comparator): Referral to a center-based cardiac rehabilitation program (standard of care).
  Interventions: Behavioral: Referral to home-based cardiac rehab

INTERVENTIONS:
Behavioral: Referral to home-based cardiac rehab — Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
  Arms: Center-based
Behavioral: Referral to center-based cardiac rehab — Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
  Arms: Home-based

SUMMARY:
The long-term goal of this research is to improve patient-centered outcomes in patients with coronary heart disease (CHD), the leading cause of death in the world. Exercise-based cardiac rehabilitation (CR) programs decrease mortality and improve quality of life in patients with CHD. Published guidelines recommend exercise-based CR following hospitalization for myocardial infarction, coronary artery bypass grafting, or percutaneous coronary revascularization.

Despite these compelling benefits, CR programs are vastly underutilized, with less than a third of eligible patients participating. One promising solution is greater implementation of home-based CR. Both home and center-based CR programs have equal benefits on cardiovascular risk factors and quality of life. However, similar efficacy does not necessarily translate into similar effectiveness. If patients are more likely to participate in home- vs. center-based therapy, then greater participation could lead to greater clinical effectiveness. We are therefore conducting a quasi-experimental, controlled trial at two VA medical centers to determine the comparative effectiveness of referral to home- vs. center-based CR in patients with CHD.

Aim 1: Determine whether automatic referral to home- vs. center-based CR increases patient participation in CR after hospitalization for myocardial infarction or coronary revascularization.

Aim 2: Among patients who choose to participate in CR, compare the effectiveness of home- vs. center-based CR on six-minute walk distance, quality of life, and healthcare expenditures.

Aim 3: Determine whether the effects of home vs. center-based CR differ by age, gender, race, ethnicity, employment, socioeconomic status, social support, comorbid conditions, or patient preference.

Results from this study will (a) help policy makers determine the effect of covering home CR on healthcare expenditures in patients with CHD; (b) help providers understand the potential benefits and harms of home- vs. center-based CR; and (c) help patients answer questions like, "Given my personal circumstances and preferences, which of these options will improve the outcomes most important to me".

DETAILED DESCRIPTION:
The long-term goal of this research is to improve patient-centered outcomes in patients with coronary heart disease (CHD). CHD is the leading cause of death in the world. Exercise-based cardiac rehabilitation (CR) programs decrease mortality and improve quality of life in patients with CHD. Published guidelines recommend exercise-based CR following hospitalization for myocardial infarction, coronary artery bypass grafting, or percutaneous coronary revascularization, and referral to CR is one of nine performance measures established by the American Heart Association and American College of Cardiology for patients with CHD.

Despite these compelling benefits, CR programs are vastly underutilized, with less than a third of eligible patients participating. The largest barrier to patient participation is that CR must be provided in a physician's office or hospital setting to qualify for reimbursement. For this reason, virtually all existing CR programs require that the patient travel to a CR center 3 times per week for 12 to 36 weeks. Unfortunately, many Americans live too far from a CR center to enroll, and even when nearby programs are available, many patients do not have the time, flexibility, transportation, social support, and/or financial resources to attend.

One promising solution to the problem of CR under-utilization is greater implementation of home-based CR. Both home and center-based CR programs have equal benefits on cardiovascular risk factors and quality of life. However, similar efficacy does not necessarily translate into similar effectiveness. If patients are more likely to participate in home- vs. center-based therapy, then greater participation could lead to greater clinical effectiveness. We are therefore conducting a quasi-experimental, controlled trial at two VA medical centers to determine the comparative effectiveness of referral to home- vs. center-based CR in patients with CHD.

Aim 1: Determine whether automatic referral to home- vs. center-based CR increases patient participation in CR after hospitalization for myocardial infarction or coronary revascularization.

Aim 2: Among patients who choose to participate in CR, compare the effectiveness of home- vs. centerbased CR on six-minute walk distance, quality of life, and healthcare expenditures.

Aim 3: Determine whether the effects of home vs. center-based CR differ by age, gender, race, ethnicity, employment, socioeconomic status, social support, comorbid conditions, or patient preference.

Results from this study will (a) help policy makers determine the effect of covering home CR on healthcare expenditures in patients with CHD; (b) help providers understand the potential benefits and harms of home- vs. center-based CR; and (c) help patients answer questions like, "Given my personal circumstances and preferences, which of these options will improve the outcomes most important to me.

ELIGIBILITY:
Inclusion Criteria:

Post MI, CABG, or PCI Able to speak, read and write in english

Exclusion Criteria:

Class IV CHF Unstable Angina Complex Ventricular Arrythmias EF <35% without AICD AICD candidate Resting SBP >200mmHG Resting DBP>110mmHG Cognitive Impairment by MoCA Score <26 Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1154 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Whooley, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Schopfer DW, Whooley MA, Allsup K, Pabst M, Shen H, Tarasovsky G, Duvernoy CS, Forman DE. Effects of Home-Based Cardiac Rehabilitation on Time to Enrollment and Functional Status in Patients With Ischemic Heart Disease. J Am Heart Assoc. 2020 Oct 20;9(19):e016456. doi: 10.1161/JAHA.120.016456. Epub 2020 Sep 21. PMID 32954885

RESULTS

PARTICIPANT FLOW:
Groups:
- Referral to Home-based Cardiac Rehabilitation: Referral to home-based cardiac rehabilitation (intervention): Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
- Referral to Center-based Cardiac Rehabilitation: Referral to center-based cardiac rehabilitation (standard of care): Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
Period: Overall Study
Arm/Group | Referral to Home-based Cardiac Rehabilitation | Referral to Center-based Cardiac Rehabilitation
Started | 557 | 597
Completed | 557 | 597
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population was as depicted in Participant Flow.
Groups:
- Home-based: Referral to home-based cardiac rehabilitation (intervention): Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
- Center-based: Referral to center-based cardiac rehabilitation (standard of care): Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
- Total: Total of all reporting groups
Arm/Group | Home-based | Center-based | Total
Number analyzed (Participants) | 557 | 597 | 1154
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years), integer
  years | 67 (9) | 66 (10) | 66.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 550 | 587 | 1137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 378 | 420 | 798
  Black | 41 | 40 | 81
  Asian | 16 | 3 | 19
  Hispanic/Latino | 51 | 4 | 55
  Missing data | 71 | 130 | 201
Region of Enrollment [Number; unit: participants]
  United States | 557 | 597 | 1154

OUTCOME MEASURES:

1. Primary Outcome: Participation in Cardiac Rehabilitation
Description: Number of eligible patients who participated in at least one cardiac rehabilitation exercise session.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- Referral to Home-based Cardiac Rehabilitation: Referral to a home-based cardiac rehabilitation program (intervention).
  Referral to home-based cardiac rehabilitation: Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
- Referral to Center-based Cardiac Rehabilitation: Referral to a center-based cardiac rehabilitation program (standard of care).
  Referral to center-based cardiac rehabilitation: Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
Arm/Group | Referral to Home-based Cardiac Rehabilitation | Referral to Center-based Cardiac Rehabilitation
Number analyzed (Participants) | 557 | 597
Participants | 231 | 252
Statistical Analysis 1: Comparison: Referral to Home-based Cardiac Rehabilitation vs Referral to Center-based Cardiac Rehabilitation; Null hypothesis = no difference in proportion of patients who participate in cardiac rehab after referral to home-based vs. facility-based programs; Test type: Equivalence — This analysis compared the proportion of eligible patients who participated in cardiac rehab after referral to home-based vs. referral to center-based programs; p = 0.80, Chi-squared; Risk Ratio (RR) = 0.98

2. Other Pre Specified Outcome: Change in Distance Completed on 6-minute Walk Test
Description: Baseline to 3-month change in 6-minute walk test distance (feet) among subjects who participated in home-based vs. center-based cardiac rehab.
Time Frame: 3 months
Population: This analysis compared 3-month change in 6-minute walk test distance among subjects who participated in home-based vs. center-based cardiac rehab. Data from participants who completed the 3 month follow up visit are presented.
Measure: Median (Inter-Quartile Range); unit: feet
Groups:
- Home-based Cardiac Rehabilitation Participants: Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
- Center-based Cardiac Rehabilitation Participants: Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
Arm/Group | Home-based Cardiac Rehabilitation Participants | Center-based Cardiac Rehabilitation Participants
Number analyzed (Participants) | 86 | 93
feet | 324 [160 to 544] | 128 [20 to 226]
Statistical Analysis 1: Comparison: Home-based Cardiac Rehabilitation Participants vs Center-based Cardiac Rehabilitation Participants; Null hypothesis: 3-month change in 6MWT distance is not inferior among participants enrolled in home-based vs. facility-based cardiac rehab; Test type: Non-Inferiority — This analysis compared Baseline to 3-month change in 6-minute walk test distance among subjects who participated in home-based cardiac rehab vs. subjects who participated in center-based cardiac rehab; p < 0.001, Wilcoxon (Mann-Whitney) — This comparison was unadjusted; Median Difference (Final Values) = 196

3. Other Pre Specified Outcome: Change in Distance Completed on 6-minute Walk Test
Description: Baseline to 6-month change in 6-minute walk test distance (feet) among patients who participated in home-based vs. center-based cardiac rehab.
Time Frame: 6 months
Population: This analysis compares 6-month change in 6-minute walk test distance (feet) among patients who participated in home-based cardiac rehab vs. patients who participated in center-based cardiac rehab.
Measure: Median (Inter-Quartile Range); unit: feet
Groups:
- Referral to Home-based Cardiac Rehab: Referral to a home-based cardiac rehabilitation program (intervention).
  Referral to center-based cardiac rehab: Center-based cardiac rehab is a health center-based cardiac rehabilitation program that involves counseling in healthy heart behaviors and exercise delivered in a clinical setting.
- Referral to Center-based Cardiac Rehab: Referral to a center-based cardiac rehabilitation program (standard of care).
  Referral to home-based cardiac rehab: Home-based cardiac rehab is a 12 week, home-based lifestyle intervention that includes counseling regarding heart healthy lifestyle changes.
Arm/Group | Referral to Home-based Cardiac Rehab | Referral to Center-based Cardiac Rehab
Number analyzed (Participants) | 33 | 70
feet | 315 [60 to 544] | 156 [56 to 305]
Statistical Analysis 1: Comparison: Referral to Home-based Cardiac Rehab vs Referral to Center-based Cardiac Rehab; Null hypothesis: 6-month change in 6MWT distance is not inferior among participants enrolled in home-based vs. facility-based cardiac rehab; Test type: Non-Inferiority — This analysis compared 6-month change in 6-minute walk test distance among subjects who participated in home-based vs. center-based cardiac rehab; p = 0.03, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 159

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event reporting data was recorded for participants who enrolled in cardiac rehab (231 home-based and 252 facility-based).
Arm/Group | Referral to Home-based Cardiac Rehabilitation | Referral to Center-based Cardiac Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/252
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/252
Other Adverse Events (participants affected / at risk) | 0/231 | 0/252

LIMITATIONS AND CAVEATS:
CR referral process differed across sites: 90% of eligible patients were referred at the San Francisco (home-based CR) site, whereas 56% of eligible patients were referred at the Ann Arbor and Pittsburgh (center-based CR) sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02105246/Prot_SAP_001.pdf